CLINICAL TRIAL: NCT00981695
Title: An Open Randomized Phase I/II Study Evaluating Safety and Immunogenicity of a Candidate HIV-1 Vaccine, MVA.HIVA, Administered to Healthy Infants Born to HIV-1-infected Mothers
Brief Title: Safety and Immunogenicity Study of Candidate HIV-1 Vaccine Given to Healthy Infants Born to HIV-1-infected Mothers
Acronym: PedVacc002
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Council (Other Government)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Tomas Hanke, Medical Research Council, UK
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: PV002
Record Dates: First submitted 2009-09-21; First posted 2009-09-22 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2009-09

CONDITIONS: HIV-1; HIV Infections
Keywords: HIV; Vaccine; MVA; PMTCT; HIV preventive vaccine; HIV seronegativity
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vaccinees (Experimental): 18 breast-fed and 18 formula-fed infants at the age of 20 weeks
  Interventions: Biological: MVA.HIVA
- Controls (No Intervention): 18 breast-fed and 18 formula-fed infants at the age of 20 weeks

INTERVENTIONS:
Biological: MVA.HIVA — 1 dose of 5 x 10^7 pfu of MVA.HIVA administered intramuscularly
  Arms: Vaccinees

SUMMARY:
Objectives:

Primary: Safety and immunogenicity of MVA.HIVA vaccine in 20-week-old healthy Kenyan infants born to HIV-1-infected mothers.

Secondary:

* HIV-1 immunogenicity comparison between MVA.HIVA and age-matched unvaccinated control arms in each cohort (breastfeeding or formula feeding)
* HIV-1 immunogenicity comparison between breastfeeding and formula feeding infants receiving MVA.HIVA
* HIV-1 immunogenicity comparison between breastfeeding and formula feeding infants in the age-matched unvaccinated control group
* Comparison of responses to certain Kenyan Extended Programme on Immunization (KEPI) vaccines (OPV, DTP, HBV, and HiB) between MVA.HIVA versus age-matched unvaccinated controls in each cohort, between breast versus formula feeding infants in the age-matched unvaccinated control group, and between breast versus formula infants receiving MVA.HIVA
* Comparison of immune activation and phenotypic profile of lymphocytes between breast and formula feeding infants in each cohort (MVA.HIVA and age-matched unvaccinated control)
* Build capacity for Infant HIV-1 Vaccine Clinical Trials Centre in Nairobi, Kenya.

ELIGIBILITY:
Infant Inclusion Criteria

* Healthy infants
* < 3 days of age (day of birth = Day 0) at enrolment
* Birth weight > 2500 grams
* Born to an eligible woman
* Written informed consent by parent

Infant Exclusion Criteria

* HIV infection, as determined by a filter paper and/or RNA test prior to vaccination.
* Participation in any other HIV-1 vaccine or drug trial.
* Failure to receive all standard KEPI immunizations according to national immunization programme.
* Weight for age z-scores outside of 2 standard deviations of normal at the time of vaccination.
* Acute disease at the time of vaccination (acute disease is defined as the presence of a moderate or severe illness with or without fever). All vaccines can be administered to persons with a minor illness such as diarrhoea, mild upper respiratory tract infection with or without low-grade febrile illness, i.e., temperature of <37.5 °C).
* Axillary temperature of ≥ 37.5 °C at the time of vaccination.
* Any clinically significant abnormal finding on screening from biochemistry or haematology by the time of vaccination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g., egg products.
* Presence of any underlying disease that compromises the diagnosis and evaluation of response to the vaccine.
* Any other on-going chronic illness requiring hospital specialist supervision.
* Administration of immunoglobulins and/or any blood products within one month preceding the planned administration of the vaccine candidate.
* Any history of anaphylaxis in reaction to vaccination.
* Research Physician's assessment of lack of willingness by parents to participate and comply with all requirements of the protocol, or identification of any factor felt to significantly increase the infant's risk of suffering an adverse outcome.
* Likelihood of travel away from the study area.

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-07 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
For safety and reactogenicity: Actively and passively collected data on adverse events. | Up to 28 weeks after vaccination

SECONDARY OUTCOMES:
For immunogenicity to KEPI vaccines: Antibody levels to specific vaccines as measured by ELISA. | 1 week before and 1 week after vaccination
For immunogenicity to MVA.HIVA: Frequency of IFN-γ-producing cells determined in an ELISPOT assay after overnight stimulation with a pool of HIVA-derived peptides. | Up to 24 weeks after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Hanke, Study Director — Medical Research Council; Walter Jaoko, Principal Investigator — University of Nairobi; Grace John-Stewart, Principal Investigator — University of Washington; Marie Reilly, Principal Investigator — Karolinska Institutet
Locations (1):
- Kenyatta National Hospital, Nairobi, Kenya

REFERENCES:
- [Derived] Njuguna IN, Ambler G, Reilly M, Ondondo B, Kanyugo M, Lohman-Payne B, Gichuhi C, Borthwick N, Black A, Mehedi SR, Sun J, Maleche-Obimbo E, Chohan B, John-Stewart GC, Jaoko W, Hanke T. PedVacc 002: a phase I/II randomized clinical trial of MVA.HIVA vaccine administered to infants born to human immunodeficiency virus type 1-positive mothers in Nairobi. Vaccine. 2014 Oct 7;32(44):5801-8. doi: 10.1016/j.vaccine.2014.08.034. Epub 2014 Aug 27. PMID 25173484